CLINICAL TRIAL: NCT04130646
Title: Combining Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) With Transcranial Magnetic Stimulation (TMS) to Enhance Cortical Excitability
Brief Title: Noninvasive VNS to Facilitate Excitability in Motor Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00089851
Record Dates: First submitted 2019-09-30; First posted 2019-10-17 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Stroke Sequelae; Motor Activity
Keywords: stroke; recovery; TMS; VNS; motor; motor cortex
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TMS combined with taVNS (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation; Device: transcutaneous auricular vagus nerve stimulation (taVNS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — transcranial magnetic stimulation delivers magnetic pulses to the brain through the scalp/skull
Device: transcutaneous auricular vagus nerve stimulation (taVNS) — non-invasive vagus nerve stimulation delivers electricity to the ear

SUMMARY:
Transcranial Magnetic Stimulation (TMS) positively influences motor rehabilitation in stroke recovery. Transcutaneous auricular vagus nerve stimulation (taVNS) has shown effects on cortical plasticity. We investigate whether combination of TMS and taVNS is more effective at motor cortex excitability than either modality alone.

DETAILED DESCRIPTION:
The investigators aim to determine the effects of taVNS on motor cortex excitability. The hypothesis is that taVNS alone (sham rTMS + active taVNS) will induce increases in motor cortex excitability (post-stimulation compared to baseline). The investigators expect these changes will be of a lesser magnitude than those of TMS alone (active rTMS + sham taVNS) due to the indirect mechanistic approach of taVNS. Another aim is to determine whether taVNS-paired TMS is more effective at inducing cortical excitability than TMS alone, as it is hypothesized that pairing two forms of neuromodulation (active rTMS + active taVNS) will increase TMS-induced cortical excitability in the motor cortex when compared to single modality approaches (active rTMS + sham taVNS; sham rTMS + active taVNS). Furthermore, it is expected that this increase is timing sensitive, and the paired approach will induce larger TMS-induced cortical excitability compared to unpaired neuromodulation (active taVNS + active taVNS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* endorsing good health

Exclusion Criteria:

* no TMS-induced motor cortex excitability changes in response to 20Hz motor cortex rTMS
* active psychiatric or neurological disorders
* history of CNS disease, concussion, overnight hospitalization, or other neurologic sequelae, tumors, seizures, frequent or severe headaches
* metal implanted above the neck
* currently taking seizure reducing medications
* currently taking psychotropic medications
* any psychotropic medication taken within 5 half-lives of procedure time
* abuse or dependence of drugs (excluding nicotine and caffeine)
* currently taking medications that lower the seizure threshold
* taking any of the stimulants, thyroid medication, or steroids
* implanted devices/ferrous metal of any kind
* history of seizure or seizure disorder
* inability to determine motor threshold.
* Pregnant females and children under the age of 18 will be excluded for safety reasons
* No vulnerable populations or special classes of subjects will be considered for participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2024-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data except through peer-review.

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS and taVNS: Transcranial Magnetic Stimulation: transcranial magnetic stimulation delivers magnetic pulses to the brain through the scalp/skull
  transcutaneous auricular vagus nerve stimulation (taVNS): non-invasive vagus nerve stimulation delivers electricity to the ear
Period: Overall Study
Arm/Group | TMS and taVNS
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 4 Separate Visits of TMS/taVNS: Transcranial Magnetic Stimulation: transcranial magnetic stimulation delivers magnetic pulses to the brain through the scalp/skull
  transcutaneous auricular vagus nerve stimulation (taVNS): non-invasive vagus nerve stimulation delivers electricity to the ear
Arm/Group | 4 Separate Visits of TMS/taVNS
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  Age 18-65 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-hispanic | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety of Combined taVNS and TMS
Description: We will monitor and record adverse events of combined taVNS TMS intervention.
Time Frame: every 10 minutes following for 30 minutes
Population: The population was analyzed for safety. The number of participants with an adverse event was recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | TMS and taVNS
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 8 months
Description: There are no adverse events reported in this study.
Arm/Group | TMS Combined With taVNS
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/46/NCT04130646/Prot_SAP_002.pdf
  • Informed Consent Form (2020-06-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT04130646/ICF_000.pdf